CLINICAL TRIAL: NCT04378101
Title: Eating Disorders Genetics Initiative (EDGI)
Brief Title: Eating Disorders Genetics Initiative
Acronym: EDGI
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Otago (Other); University of Aarhus (Other); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1378; R01MH120170 (NIH)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-04

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
Keywords: Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Participants from the United States, Australia, and New Zealand will be asked to submit a saliva sample using standard industry collection tubes. DNA will be isolated from these samples.
  DNA will be isolated from blood spots obtained at birth from participants in Denmark.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anorexia Nervosa Case: Participants in this group have a life-time history of anorexia nervosa as determined by an algorithm applied to their responses to an eating disorders screening questionnaire (ED100K) that is based on the Structured Clinical Interview for Axis 1 Disorders.
  Interventions: Other: Eating disorder diagnosis group
- Bulimia Nervosa Case: Participants in this group have a life-time history of bulimia nervosa as determined by an algorithm applied to their responses to an eating disorders screening questionnaire (ED100K) that is based on the Structured Clinical Interview for Axis 1 Disorders. These participants do not have a history of anorexia nervosa.
  Interventions: Other: Eating disorder diagnosis group
- Binge-Eating Disorder Case: Participants in this group have a life-time history of binge-eating disorder as determined by an algorithm applied to their responses to an eating disorders screening questionnaire (ED100K) that is based on the Structured Clinical Interview for Axis 1 Disorders. These participants do not have a history of anorexia nervosa or bulimia nervosa.
  Interventions: Other: Eating disorder diagnosis group
- Control: Participants in this group have no history of disordered eating behaviors as determined by an algorithm applied to their responses to an eating disorders screening questionnaire (ED100K) that is based on the Structured Clinical Interview for Axis 1 Disorders.
  Interventions: Other: Eating disorder diagnosis group

INTERVENTIONS:
Other: Eating disorder diagnosis group — This is an observational study, no active intervention is applied. Participants are assigned to an eating disorder diagnosis group based on their lifetime history of disordered eating behaviors and symptoms.

SUMMARY:
The overarching intention of the Eating Disorder Genetics Initiative (EDGI) is to lay the foundation for all future genomic discovery in eating disorders--anorexia nervosa (AN), bulimia nervosa (BN), and binge-eating disorder (BED)--by exploring both genetic and behavioral factors. To do this, information will be collected from 4000 people who have provided DNA samples for the Anorexia Nervosa Genetics Initiative (ANGI) and the same information and DNA will be collected from an additional 16,000 people. The goal is to better understand eating disorders and how they relate to each other so that better treatments can be developed.

ELIGIBILITY:
Inclusion Criteria:

* A lifetime history of anorexia nervosa, bulimia nervosa, binge-eating disorder, or no history of any disordered eating behavior
* Age 15-99 years

Exclusion Criteria:

* History of subthreshold disordered eating behaviors

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Interested individuals from the United States, Australia, and New Zealand who meet criteria may participate within their respective country.
Sampling Method: Non-Probability Sample
Enrollment: 17991 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants Identified with an Eating Disorder Diagnosis by Category | Baseline
  The ED100K is a web-based diagnostic questionnaire, based on the Structured Clinical Interview for Axis 1 Disorders, that applies algorithms to participant responses. The number of participants with each diagnosis (AN, BN, BED, and control) will be reported.
Age of eating disorder onset | Baseline
  Age of eating disorder onset will be considered as the age of first eating disorder symptom as self-reported in the ED100K questionnaire (ED100K). Age of onset will be reported for each eating disorder group.

SECONDARY OUTCOMES:
Current eating disorder self-report total sum scores | Baseline
  Current eating disorder symptoms will be determined by self-report responses on the Eating Disorder Examination Questionnaire (EDEQ). Items ask about eating disorder symptoms over the past 28 days. There are four subscales of the EDEQ--Restraint, Eating Concern, Shape Concern, and Weight Concern--with scores for each ranging from 0-6. Subscales are averaged to compute a total score. Higher scores indicate more eating disorder pathology. Total and subscale sores will be reported to each eating disorder group.
Eating disorder-related quality of life scores | Baseline
  Eating disorder quality of life will be measured with the Eating Disorder Quality of Life (EDQL) self-report questionnaire. The EDQL asks 25 items about the psychological, physical, financial, and work/school impact of an eating disorder over the past 30 days. Items are scored never (0), rarely (1), sometimes (2), often (3), or always (4). Items are summed for a total score ranging from 0-100, representing the overall impact of an eating disorder on life quality. Higher scores indicate a more significant impact of the eating disorder on life quality. Scores will be reported for each eating disorder group.
Health-related quality of life scores | Baseline
  Quality of life will be measured with the Short Form Health Survey 12 (SF-12) self-report questionnaire. The SF-12 asks 12 items assessing physical and mental health scores range from 0 to 100, with higher scores indicating better quality of life. Scores will be reported for each eating disorder group and for controls.
Current depressive symptoms sum score | Baseline
  Current depressive symptoms will be measured using the Patient Health Questionnaire (PHQ). The PHQ asks 9 items about symptoms of depression over the past 2 weeks. Response options range from 0 (not at all) to 3 (nearly every day). Items are summed for a total score, ranging between 0-27 with higher scores indicating more depressive symptoms. Scores will be reported for each eating disorder group and for controls.
Prevalence of life-time history of major depression | Baseline
  The prevalence of a history of major depression will be compared between eating disorder groups. Participants will complete a self-report questionnaire with items linked to the diagnostic criteria for major depression. Those individuals who indicate the presence of all the criterion required for a major depression diagnosis will be considered to have a history of major depression. Prevalence of life-time history of major depression will be reported for each eating disorder group and for controls.
Current anxiety symptoms sum scores | Baseline
  Current anxiety symptoms will be measured using the Generalized Anxiety Disorder 7 (GAD7) self report questionnaire. GAD7 is a questionnaire for screening and severity measuring of generalized anxiety disorder. GAD7 consists of a total score for the seven items ranging from 0 to 21. Higher scores indicate higher levels of generalized anxiety. Scores will be reported for each eating disorder group and for controls.
Prevalence of generalized anxiety disorder | Baseline
  The prevalence of a history of a generalized anxiety disorder will be compared between eating disorder groups. Participants will complete a self-report questionnaire with items linked to the diagnostic criteria for an anxiety disorder. Those individuals who indicate the presence of all the criterion required for generalized anxiety disorder diagnosis will be considered to have a history of generalized anxiety disorder. The prevalence of generalized anxiety disorder will be reported for each eating disorder group and for controls.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Bulik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- University of North Carolina, Chapel Hill, North Carolina, United States
- QIMR Berghofer, Brisbane, Queensland, Australia
- University of Otago, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and scripts will be made available to the general scientific community at the conclusion of the investigation. Specifically, phenotype data will be submitted to the database of Genotypes and Phenotypes (dbGaP) and National Institute of Mental Health Repository & Genetics Resource (NRGR) and genotype data to dbGaP.
Supporting Information: Study Protocol
Time Frame: Assessment phenotype data will be submitted within 6 months after the end of the study. Genotype data will be submitted after the first set of analyses with these data are complete. All data will be available as long as the repositories maintain the datasets (indefinitely).
Access Criteria: The databases are controlled-access meaning that individuals who wish to have access to the data must apply to the respective repository and meet all of their criteria.
URL: https://nda.nih.gov/nda/access-data-info.html

REFERENCES:
- [Derived] Watson HJ, Schaumberg K, Thornton LM, Kennedy HL, Ong SH, Roche P, Barnhart WR, Pauley-Gadd SB, Costello K, Flatt RE, Birgegard A, Dinkler L, Abbaspour A, Mantilla EF, Monell E, Frans EM, Barakat S, Pettie MA, Parker R, Maguire S, Jordan J, Kennedy MA, Bulik CM. Maladaptive Exercise in People With a Lifetime History of Eating Disorders: A Multicountry Observational Study. Int J Eat Disord. 2026 Jan;59(1):190-204. doi: 10.1002/eat.24563. Epub 2025 Oct 20. PMID 41115789
- [Derived] Bulik CM, Thornton LM, Parker R, Kennedy H, Baker JH, MacDermod C, Guintivano J, Cleland L, Miller AL, Harper L, Larsen JT, Yilmaz Z, Grove J, Sullivan PF, Petersen LV, Jordan J, Kennedy MA, Martin NG. The Eating Disorders Genetics Initiative (EDGI): study protocol. BMC Psychiatry. 2021 May 4;21(1):234. doi: 10.1186/s12888-021-03212-3. PMID 33947359